CLINICAL TRIAL: NCT01974401
Title: Effect of Using Supragingival Irrigators Containing Chlorhexidine on Oral Health in Patients With Blood Dyscrasia
Brief Title: Effect of Supragingival Irrigators Containing Chlorhexidine on Oral Health in Blood Dyscrasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Pegah Mosannen Mozafari, assistant professor of oral medicine, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 89462
Record Dates: First submitted 2013-10-26; First posted 2013-11-01 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Severe Neutropenia; Thrombocytopenia; Chemotherapy; Blood Dyscrasia Patients
Keywords: oral irrigator; leukemia; blood dyscrasia; Oral Health Index Simplified (OHI-S); supra gingival irrigator
MeSH Terms: conditions — Neutropenia; Thrombocytopenia; Leukemia; Hematologic Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- water jet irrigator (Active Comparator): patients used supra-gingival irrigators as an oral health measure
  Interventions: Device: supragingival irrigators containing chlorhexidine
- control group (No Intervention): patients in this group received routine oral health care protocols.

INTERVENTIONS:
Device: supragingival irrigators containing chlorhexidine — patients received irrigation by oxyjet supra gingival irrigators containing chlorhexidine for at least 3 minutes for all dentulous regions of jaws which was performed by researchers once daily.
  Other Names: Oral-B Braun Oxyjet irrigators
  Arms: water jet irrigator

SUMMARY:
in this study , effectiveness of supragingival irrigators containing chlorhexidine is compared with routine oral health measures in patients with blood dyscrasia whom can not use effective oral health measures(e.g brushing ) due to their systemic condition(e,g,neutropenia ,thrombocytopenia,..)

DETAILED DESCRIPTION:
Since some patients with hematologic malignancies cannot brush effectively and are at increased risk of bleeding and infection due to severe neutropenia and thrombocytopenia we want to access whether a none invasive method ( water jet systems containing chlorhexidine ) Can help this patients to get better oral health indexes in comparison with routine oral health measures in these type of patients.

ELIGIBILITY:
Inclusion Criteria:

patients with a blood dyscrasia, severe neutropenia and thrombocytopenia, absence of periodontitis, absence of any oral mucosal lesion in onset of study, patient consent

Exclusion Criteria:

diabetes mellitus, observation of any side effect (resulted from the device), severe oral mucositis in intervention group(grade 3 and4 WHO), edentulousness, intolerance of device in severely malaise patients, patient death

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2011-03 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
improvement in oral health status | 3 weeks
  improvement of oral health was measured by oral health index simplified(OHI-S)

SECONDARY OUTCOMES:
incidence of oral mucositis | 3 weeks
  incidence of mucositis due to Who criteria explored by clinical examination

CONTACTS AND LOCATIONS:
Overall Officials: Pegah Mosannen Mozafari, assistant professor, Study Director — Oral and maxilloifacial diseases research center of Mashhad university of medical sciences
Locations (1):
- Oral Medicine Department of Mashhad dental School,Oral and Maxillofacial diseases research center, Mashhad, Khorasan Razavi, Iran